CLINICAL TRIAL: NCT06019533
Title: A Multicentre, Single Arm Trial on Contraceptive Efficacy, Safety and Tolerability of LVDS (Levonorgestrel Vaginal Delivery System) During 13 Cycles
Brief Title: A Trial on Contraceptive Efficacy, Safety and Tolerability of LVDS (Levonorgestrel Vaginal Delivery System) During 13 Cycles
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chemo Research (Industry)
Responsible Party: Sponsor
Organization: Insud Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: LR-301
Record Dates: First submitted 2023-08-25; First posted 2023-08-31 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Contraception

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- LVDS (Experimental)
  Interventions: Combination Product: LVDS

INTERVENTIONS:
Combination Product: LVDS — Levonorgestrel Vaginal Delivery System

SUMMARY:
Multicentre, single arm phase III trial to assess the pearl index of LVDS. The trial lasts 13 cycles.The assessments include (but are not limited to) recording demographic data, pregnancy tests, gynaecological examinations, laboratory tests and a quality of life questionnaire. Adolescents will undergo DXA scans to measure bone mineral density (at selected sites only). The women will be provided with an e-diary app for their smartphone, to record IP use and vaginal bleeding.

ELIGIBILITY:
Inclusion Criteria:

* At Visit 1a, subjects must meet ALL of the following criteria:

  1. Sexually active, postmenarcheal and premenopausal female subjects at risk of pregnancy including breastfeeding women.
  2. Women who either

     1. have never used hormonal contraceptives before consent/assent (naïve users), or
     2. have used hormonal contraceptives in the past, but have had a hormonal contraceptive-free period before consent/assent and a full menstrual cycle during the drug-free period (previous users) or
     3. directly switch from another hormonal contraceptive (switchers).
  3. Only for subjects who were not pregnant and did not use hormonal contraception during the last 6 months before consent/assent:

Regular cycles (i.e. cycle length between 24 and 35 days) during the last 6 months.

Exclusion Criteria:

1. Pregnancy or wish of pregnancy.
2. Subject is known to or suspected of not being able to comply with the trial protocol, the use of the trial medication or the use of the trial diary.
3. History of infertility.
4. Known bleeding disorder or history of unexplained bleeding or bruising within the last 12 months prior to V1a.
5. Unexplained amenorrhoea.
6. Abnormal finding on pelvic, breast or ultrasound examination that in the investigator's opinion contraindicates participation in the trial.

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 750 (Estimated)
Dates: Start 2023-08-09 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Pearl Index | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- LR-301/, Móstoles, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No